CLINICAL TRIAL: NCT05263544
Title: Evaluation of Uterine Anatomical Flexion Degree ( Uterocervical Angle) in Cases With and Without Intrauterine Device (IUD) Dislocation
Brief Title: Uterine Anatomical Flexion Degree ( Uterocervical Angle) and Intrauterine Device (IUD) Dislocation
Status: Completed | Type: Observational
Sponsor: Gaziosmanpasa Research and Education Hospital (Other Government)
Responsible Party: Principal Investigator, Fatma Ketenci Gencer, MD, Principal investigator, Gaziosmanpasa Research and Education Hospital
Other Study IDs: GaziosmanpasaTREHg
Record Dates: First submitted 2022-02-03; First posted 2022-03-02 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2023-06

CONDITIONS: Contraception; Intrauterine Device Dislocation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with displaced IUD
  Interventions: Other: measuring uterocervical angle and uterine dimensions
- Patients without displaced IUD
  Interventions: Other: measuring uterocervical angle and uterine dimensions

INTERVENTIONS:
Other: measuring uterocervical angle and uterine dimensions — in both groups with and without displaced IUD, uterus size, uterine width, cervical canal length, endometrial canal length, endometrial canal width, and the angle at the intersection of the imaginary lines corresponding to the middle of the endometrium and cervical canal, which can be detected by transvaginal ultrasound will be measured

SUMMARY:
Investigators want to find numerical determination of the degree of anatomical anterior or posterior flexion of the uterus (uterocervical angle) at the intersection of both lines using a protractor, provided that straight lines are drawn from the middle of the cervical canal and the middle of the endometrial canal in cases where the intrauterine device is found to have dislocated and and cases with no dislocation. Investigators will also measure uterus size, uterine width, cervical canal length, endometrial canal length, endometrial canal width and compare the results in both groups.

DETAILED DESCRIPTION:
IUD (intrauterine device) is one of the most preferred birth control methods in our country and in the world, and this usage rate is approximately 23% in the world. In our country, this rate is around 17%. The high chance of success, ease of use and long-term effectiveness can be counted among the reasons for preference.Currently used IUD is a 'T' shaped, has a 380 mm copper surface and its arms open at the widest part of the endometrium (TCu380A), thereby preventing it from slipping back. Undesirable effects include pelvic pain, dysmenorrhea, heavy menstrual bleeding, malposition/dislocation. Malposition/dislocation occurs in approximately 10% of patients. Malposition/dislocation of the IUD may be associated with excessive menstrual bleeding, or the IUD may be displaced without any symptoms. Malposition/dislocation can be classified as expulsion, burial, displacement, or perforation. Expulsion is defined as partial or complete protrusion of the cervical canal, and displacement is defined as rotation of the IUD or its displacement towards the lower segments. At the same time, IUD may be embedded in the myometrium to such an extent that it does not reach the serosa of the myometrium, while it may puncture the serosa and cause perforation may occur. TCu380A devices have a 6% risk of expulsion in the first 1 year. Displacement or slippage of the IUD reduces the effectiveness of the IUD and may cause expulsion. Therefore, being able to predict that the IUD will not slip is very important in terms of preventing unwanted pregnancies. In our study, in both groups with and without displaced IUD, uterus size, uterine width, cervical canal length, endometrial canal length, endometrial canal width, and the angle at the intersection of the imaginary lines corresponding to the middle of the endometrium and cervical canal, which can be detected by transvaginal ultrasound were measured. Investigators aimed to determine the measurements and compare the obtained data to find associated factors related to dislocation.

ELIGIBILITY:
Inclusion Criteria:

• using intrauterine device

Exclusion Criteria:

* Pelvic mass that cannot be differentially diagnosed by physical examination and imaging techniques
* Having an indication for surgical treatment
* Presence of space-occupying polyp or fibroid affecting the anatomy of the endometrium
* Presence of myoma or adenomyosis that disrupts the integrity of the myometrium
* Presence of pelvic infection
* Currently using any hormonal therapy
* History and/or presence of malignancy
* Pregnancy
* Menopause or premature ovarian failure

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: patients with and without intrauterine device displacement
Sampling Method: Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2021-06-30 (Actual); Primary Completion 2023-03-15 (Actual); Study Completion 2023-03-28 (Actual)

PRIMARY OUTCOMES:
Determination of factors associated with intrauterine device dislocation. | 6 months
  Degree of uterocervical angle (°)will be measured and assessed for association with dislocation.
Determination of factors associated with intrauterine device dislocation. | 6 months
  uterus size (mm) will be measured and assessed for association with dislocation.
Determination of factors associated with intrauterine device dislocation. | 6 months
  uterine width (mm) will be measured and assessed for association with dislocation.
Determination of factors associated with intrauterine device dislocation. | 6 months
  cervical canal length(mm) will be measured and assessed for association with dislocation.
Determination of factors associated with intrauterine device dislocation. | 6 months
  endometrial canal length (mm) will be measured and assessed for association with dislocation.
Determination of factors associated with intrauterine device dislocation. | 6 months
  endometrial canal width (mm) will be measured and assessed for association with dislocation.

CONTACTS AND LOCATIONS:
Overall Officials: Fatma Ketenci Gencer, MD, Principal Investigator — Saglik Bilimleri Universitesi
Locations (1):
- Gaziosmanpasa Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes